CLINICAL TRIAL: NCT05831488
Title: Assessing the Accuracy of Seismofit® as an Estimate of VO2 Peak in Patients With Hepato-pancreato-biliary, Colorectal, and Gastro-oesophageal Cancer
Acronym: VERVE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR5651
Record Dates: First submitted 2023-01-17; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-01

CONDITIONS: Hepato-Biliary Carcinoma in Situ Nos; Pancreatic Cancer; Colorectal Cancer; Gastric Cancer; Oesophageal Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Colorectal Neoplasms; Stomach Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non-Interventional — Non Interventional

SUMMARY:
Our study aims to assess the relationship between the Seismofit® derived VO2 peak estimate and CPET-measured VO2 peak in patients who are having CPET as part of their preoperative workup. Our aim is to establish whether Seismofit® can be considered a cheaper, less resource intensive and better tolerated alternative to the CPET, or whether it might be useful as a screening tool to efficiently identify patients with exercise intolerance who may benefit from further characterisation by CPET.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18
2. Scheduled for elective surgery for resection of HPB, colorectal or gastro-oesophageal primary or secondary cancer
3. Undergoing CPET as part of routine pre-operative investigations

Exclusion Criteria:

1. Subjects unable to give voluntary written informed consent to participate in this study
2. Diagnosis of moderate or worse stenosis or regurgitation of any cardiac valve
3. Previous aortic or mitral valve surgery, valvuloplasty or transcatheter valve implantation
4. Permanent pacemaker or cardiac resynchronisation device in situ
5. Diagnosis of severe pulmonary hypertension
6. Permanent atrial fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All HPB, gastro-oesophageal or colorectal cancer patients undergoing preoperative assessment for major surgery
Sampling Method: Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Assess the relationship between Seismofit®-estimated VO2 peak and CPET-measured VO2 peak in HPB, gastro-oesophageal or colorectal cancer patients undergoing preoperative assessment for major surgery. | End of Trial (9 months)
  Strength and direction of relationship (Pearson correlation coefficient) between Seismofit® -estimated VO2 peak and CPET-measured VO2 peak.

SECONDARY OUTCOMES:
Assess limits of agreement and bias between Seismofit®-estimated VO2 peak and CPET-measured VO2 peak | End of Trial (9 months)
  Limits of agreement and bias between Seismofit®-estimated VO2 peak and CPET-measured VO2 peak (Bland-Alman analysis)
Assess the relationship between Seismofit®-estimated VO2 peak and CPET-measured VO2 peak in each surgical subgroup: HPB, gastro-oesophageal and colorectal cancer patients. | End of Trial (9 months)
  Strength and direction of relationship (Pearson correlation coefficient) between Seismofit® -estimated VO2 peak and CPET-measured VO2 peak, as well as limits of agreement and bias (Bland-Altman analysis) in each surgical subgroup: HPB, gastro-oesophageal and colorectal cancer patients.
Assess the relationship between Seismofit® -estimated VO2 peak and other CPET derived variables: o Anaerobic Threshold (AT) o Peak Power Output (PPO) o Ventilatory equivalents for carbon dioxide (VE/VCO2) | End of Trial (9 months)
  Strength and direction of relationship (Pearson correlation coefficient) between Seismofit® -estimated VO2 peak and the CPET-measured variables of AT, PPO and VE/VCO2
Assess patient experience of the Seismofit® test using a brief measure that has been used previously in CPET research | End of Trial (9 months)
  Patient concern, comfort, and overall satisfaction of Seismofit® measurement compared with CPET.

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Marsden NHS Foundation Trust, London, United Kingdom

REFERENCES:
- [Derived] Tetlow N, Devendra P, Waiting J, Aresu M, Glover A, Rooms M, Jhanji S, Milliken D. Assessing the accuracy of Seismofit(R) as an estimate of preoperative maximal oxygen consumption in patients with hepato-pancreato-biliary, colorectal, and gastro-oesophageal cancer. BJA Open. 2025 Apr 8;14:100395. doi: 10.1016/j.bjao.2025.100395. eCollection 2025 Jun. PMID 40248106